CLINICAL TRIAL: NCT06021249
Title: Comparing the Effects of Innovative and Traditional Lung-protective Ventilation Strategies on the Occurrence of Perioperative Atelectasis and Prognosis in Elderly Patients: a Prospective, Randomized, Controlled Study
Brief Title: Comparing Innovative and Traditional Ventilation Strategies on Atelectasis and Prognosis in Elderly Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fujian Medical University Union Hospital (Other)
Collaborators: The First Affiliated Hospital of Nanchang University (Other); The First Hospital of Putian City, Putian, Fujian (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 2021MZK04KY
Record Dates: First submitted 2023-08-02; First posted 2023-09-01 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Ventilator-associated Lung Injury; Atelectasis; Postoperative Pulmonary Complications
Keywords: perioperative strategies for lung-protective ventilation; elderly patients; atelectasis; postoperative pulmonary complications; lung injury
MeSH Terms: conditions — Pulmonary Atelectasis; Lung Injury

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Group of Control (Part I experiment) (Sham Comparator): Traditional ventilation strategies
  Interventions: Procedure: Traditional ventilation strategies
- Group of traditional lung-protective ventilation (Part I experiment) (Experimental): Traditional lung-protective ventilation strategies
  Interventions: Procedure: Traditional lung-protective ventilation strategies
- Group of innovative lung-protective ventilation (Part I experiment) (Experimental): Innovative lung-protective ventilation strategies
  Interventions: Procedure: Innovative lung-protective ventilation strategies
- Group of traditional & innovative ventilation (Part I experiment) (Experimental): Traditional & innovative lung protection ventilation strategies
  Interventions: Procedure: Traditional lung-protective ventilation strategies; Procedure: Innovative lung-protective ventilation strategies
- Group of Control (Part II experiment) (Sham Comparator): 1. lung-protective ventilation；
  2. negative pressure extubation
  Interventions: Procedure: Lung-protective ventilation; Procedure: negative pressure extubation
- Group of positive pressure extubation (Part II experiment) (Experimental): 1. lung-protective ventilation；
  2. positive pressure extubation
  Interventions: Procedure: Lung-protective ventilation; Procedure: positive pressure extubation
- Group of breathing training (Part II experiment) (Experimental): 1. lung-protective ventilation；
  2. negative pressure extubation；
  3. postoperative breathing training
  Interventions: Procedure: Lung-protective ventilation; Procedure: negative pressure extubation; Procedure: postoperative breathing training
- Group of positive pressure extubation & breathing training (Part II experiment) (Experimental): 1. lung-protective ventilation；
  2. positive pressure extubation；
  3. postoperative breathing training
  Interventions: Procedure: Lung-protective ventilation; Procedure: positive pressure extubation; Procedure: postoperative breathing training

INTERVENTIONS:
Procedure: Traditional ventilation strategies — 1. Tidal volume：10ml/kg predicted body weight（PBW）；
  2. 0 cm H2O positive end expiratory pressure（PEEP）；
  3. negative pressure extubation
  Arms: Group of Control (Part I experiment)
Procedure: Traditional lung-protective ventilation strategies — 1. Tidal volume：6ml/kg PBW；
  2. 5cmH2O PEEP；
  3. Ventilator-controlled recruitment manoeuvre；
  4. CPAP；
  5. negative pressure extubation
  Arms: Group of traditional & innovative ventilation (Part I experiment); Group of traditional lung-protective ventilation (Part I experiment)
Procedure: Innovative lung-protective ventilation strategies — 1. Tidal volume：6ml/kg PBW；
  2. 5cmH2O PEEP；
  3. positive pressure extubation；
  4. postoperative breathing training
  Arms: Group of innovative lung-protective ventilation (Part I experiment); Group of traditional & innovative ventilation (Part I experiment)
Procedure: Lung-protective ventilation — 1. Tidal volume：6ml/kg PBW；
  2. 5cmH2O PEEP；
  Arms: Group of Control (Part II experiment); Group of breathing training (Part II experiment); Group of positive pressure extubation & breathing training (Part II experiment); Group of positive pressure extubation (Part II experiment)
Procedure: negative pressure extubation — The suction tube is inserted into the endotracheal tube, continuous negative pressure suction, and at the same time that the balloon is completely deflated, the suction tube, dental pad and endotracheal intubation are pulled out at the same time, and then the patient is instructed to cough independently and remove sputum.
  Arms: Group of Control (Part II experiment); Group of breathing training (Part II experiment)
Procedure: positive pressure extubation — The adjustable pressure limiting（APL）was adjusted to 30cm H2O, and after the patient breathed spontaneously until the peak airway pressure reached 30cm H2O, and after maintaining this level for 10s, the balloon was quickly cut off to remove the endotracheal tube, so that the patient had an autonomous coughing action, and then the oral sputum was removed.
  Arms: Group of positive pressure extubation & breathing training (Part II experiment); Group of positive pressure extubation (Part II experiment)
Procedure: postoperative breathing training — Inhale deeply through the nose, hold the breath for 5s, and then slowly spit out the breath through the mouth, cycle 5-6 times, and inflate the balloon. The above steps need to be performed 15 times within 24 hours after surgery.
  Arms: Group of breathing training (Part II experiment); Group of positive pressure extubation & breathing training (Part II experiment)

SUMMARY:
This study was divided into two parts, taking elderly patients undergoing general anesthesia surgery as the research subjects, through factorial design: 1. It was verified that in elderly patients undergoing general anesthesia surgery, innovative lung-protective ventilation strategies can reduce the occurrence of atelectasis and reduce the incidence of ventilator-related lung injury and postoperative pulmonary complications more than traditional lung-protective ventilation strategies; 2. On the basis of part one study proving that innovative lung-protective ventilation strategies can reduce the incidence of postoperative atelectasis and other complications in elderly patients undergoing general anesthesia surgery compared with traditional lung-protective ventilation strategies, further comparisons were made between the two factors of "positive pressure extubation" and "improved early postoperative respiratory training" in the innovative lung protective ventilation strategy, and whether there was an interaction between the two.

DETAILED DESCRIPTION:
More and more people need to undergo general anesthesia surgery at least once in the lifetime, and patients who undergo general anesthesia surgery often have postoperative pulmonary complications, and the occurrence of postoperative pulmonary complications is related to the prolongation of the patient's hospital stay and postoperative mortality. This is contrary to the current goal of rapid postoperative recovery.

The International Expert Consensus on Strategies for Pulmonary Protective Ventilation states that age > 50 years is one of the greatest risk factors for postoperative pulmonary complications. This means that even older patients with largely unimpaired preoperative lung function are more likely to develop postoperative pulmonary complications than younger patients. Therefore, the investigators set the study to elderly patients undergoing general anesthesia surgery.

The traditional lung-protective ventilation strategies commonly used to reduce atelectasis and ventilator-related lung injury during general anesthesia surgery is controversial and mixed. Based on literature review and preliminary experiments, this study focuses on extubation and post-extubation, which is a critical period of atelectasis development, combines positive pressure extubation technology with improved postoperative early breathing training, replaces the controversial continuous positive airway pressure（CPAP）support and alveolar recruitment manoeuvres in traditional lung protective ventilation strategies, and explores a new respiratory management strategy with more operability and clinical effect to reduce complications such as postoperative atelectasis in elderly patients.

This study was originally a single-center clinical study and has been registered in the Chinese Clinical Trial Registry（Registration number：ChiCTR2300071364）. It was later changed to a multi-center clinical study, so it was re-registered.

ELIGIBILITY:
Inclusion Criteria:

1. Elderly patients aged ≥ 60 years old who undergo laparoscopic abdominal surgery；
2. Body mass index（BMI） <30；
3. American society of anesthesiologists physical status classification system（ASA）:I-III；
4. When the patient inhales air before surgery, SPO2≥94%；
5. The duration of the operation is 2-7 hours, and the pneumoperitoneal pressure is 10-14mmHg.

Exclusion Criteria:

1. Patients with acute respiratory distress syndrome or pulmonary hypertension (pulmonary systolic blood pressure ≥ 40mmHg) or bronchiectasis or lung malignant tumors
2. Patients with acute respiratory infections within one month before surgery
3. Patients who have undergone cardiopulmonary surgery
4. Receiving invasive mechanical ventilation for more than 30min within 30 days before surgery
5. Patients with peak airway pressure > 35 cm H2O during intraoperative mechanical ventilation
6. Patients with severe organic lesions of the heart such as obvious heart failure and coronary heart disease
7. Patients with preoperative anemia (Hb<10g/L)
8. Patients with hypoproteinemia before surgery (albumin < 35 g/L)
9. Patients with tracheostomy and severe difficult airway
10. Patients with sleep apnea syndrome
11. Patients with intraoperative heavy bleeding (50% of the circulating blood volume is lost ≥ 3 hours)
12. Patients with mental illness, impaired consciousness and communication disorders
13. Patients who refuse to participate in this trial

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Estimated)
Dates: Start 2021-09-28 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Volume ratio of new-onset atelectasis after surgery | Pre-surgery;Approximately 24 hours after surgery
  After lung CT examination, the postoperative volume ratio of new atelectasis (new atelectasis volume/total lung volume) was calculated.

SECONDARY OUTCOMES:
postoperative pulmonary complications | Within 14 days after surgery; Within 30 days after surgery
  Diagnosis according to the US Centers for Disease Control definition of pneumonia:
  Two or more serial chest radiographs with at least one of the following (one radiograph is sufficient for patients with no underlying pulmonary or cardiac disease):
  (i) New or progressive and persistent infiltrates, (ii)consolidation, (iii) cavitation;
  AND at least one of the following:
  1. fever (>38°C) with no other recognised cause,
  2. leucopaenia (white cell count <4*10^9/ litre) or leucocytosis(white cell count >12*10^9 /litre),
  3. for adults >70 years old, altered mental status with no other recognised cause;
  AND at least two of the following:
  1. new onset of purulent sputum or change in character of sputum, or increased respiratory secretions, or increased suctioning requirements,
  2. new onset or worsening cough, or dyspnoea, or tachypnoea,
  3. rales or bronchial breath sounds,
  4. worsening gas exchange (hypoxaemia, increased oxygen requirement, increased ventilator demand).
specific indexes of ventilator-related lung injury | Pre-surgery;Immediately after the extubation;Approximately 24 hours after surgery
  Blood was drawn and centrifuged for serum ELISA to detect landmark indicators of ventilator-related lung injury
oxygenation index | Pre-surgery;20 minutes after the intubation;End of the operation;Approximately 10 minutes after the extubation;Approximately 40 minutes after the extubation;Approximately 70 minutes after the extubation;Approximately 24 hours after surgery
  Arterial blood samples are drawn for blood gas analysis

CONTACTS AND LOCATIONS:
Overall Officials: Zhongmeng Lai, Principal Investigator — Fujian Medical University Union Hospital
Locations (3):
- China (3):
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - The First Hospital of Putian, Putian, Fujian
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi

IPD SHARING:
Plan to Share IPD: Yes
In June 2024, raw data was shared through ResMan（http://www.medresman.org.cn/login.aspx）
Supporting Information: Study Protocol, ICF
Time Frame: In June 2024, raw data was shared for 6 months.
Access Criteria: Accessible to any researcher
URL: http://www.medresman.org.cn/login.aspx